CLINICAL TRIAL: NCT06532864
Title: Effects of Qigong Exercise and Mawangdui Guiding Technique on Sleep Quality in the Elderly
Brief Title: Qigong Exercise and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Huan Liu, teacher, Hunan University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022XH0111
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-07

CONDITIONS: Sleep Quality
Keywords: sleep quality; older adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to experimental and control groups. The experimental group performed Mawangdui Guided Technique exercises, which consisted of five 45-minute sessions per week for 12 weeks. The control group maintained a routine of sleep education in addition to their daily activities.
Who Masked: Outcomes Assessor
Masking Description: The investigator of the statistical analysis was unaware of the grouping of the subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Practicing Mawangdui Guidance Exersize Group (Experimental): The experimental group underwent the Mawangdui Guided Exercise, which consisted of five 45-minute sessions per week for 12 weeks.
  Interventions: Behavioral: Practice Mawangdui Guiding Technique
- Sleep Education Group (No Intervention): The control group maintained routine sleep education in addition to daily activities.

INTERVENTIONS:
Behavioral: Practice Mawangdui Guiding Technique — Nursing staff with experience in teaching Mawangdui Daoyin Exercise conducted the operation instruction on different floors. A feasibility assessment of the older adults was carried out by the nursing staff at the end of the teaching, and only after passing this assessment could the experimental part begin. The treatment group participated in five Mawangdui Daoyin Exercise sessions per week, each lasting approximately 45 minutes, and the exercises continued for 12 weeks.
  Arms: Practicing Mawangdui Guidance Exersize Group

SUMMARY:
The purpose of this study was to investigate whether 12 weeks of practicing Mawangdui Guiding Technique has an improvement effect on subjective sleep quality, objective sleep quality, and daytime fatigue in older adults in a healthcare hospital.

ELIGIBILITY:
Inclusion Criteria:

* Aged sixty years and above; continuous residence in the participating healthcare hospitals for more than six months
* Conscious, with basic visual and auditory perception, communication, and cognitive functioning
* Voluntary enrollment in this study and signing of the informed consent form.

Exclusion Criteria:

* Individuals who have suffered a sudden accident, emergency surgery, or a rapid deterioration of a long-term medical condition
* Individuals who have recently been involved in other rehabilitation activities and who play sports on a regular basis
* Individuals who are unable to participate in physical activity (e.g., patients suffering from major diseases of the liver, kidneys, heart, brain, or blood system)
* Individuals suffering from deep venous thrombosis; individuals with musculoskeletal problems with signs of limitation of movement (e.g., unsettled broken bones, pelvic fractures)
* Individuals with preexisting psychiatric conditions (such as personality disorders, psychosis, and so on); and individuals with symptoms of severe depression.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | baseline; 4 weeks; 12weeks
  The Pittsburgh Sleep Quality Index is a comprehensive sleep self-assessment tool containing 19 items. The overall total score ranges from 0-21, with the lower the overall score, the higher the quality of sleep.
Insomnia Severity Index | baseline; 4 weeks; 12weeks
  The Insomnia Severity Index(ISI) is a self-assessment tool consisting of seven items designed to assess various aspects of insomnia. Cumulative ISI scores range from 0 to 28 and are categorized as follows: 0-7 = no insomnia; 8-14 = mild insomnia; 15-21 = moderate insomnia; and 22-28 = severe insomnia.
Polysomnography | baseline; 4 weeks; 12weeks
  Polysomnography is the internationally recognized gold standard for diagnosing sleep disorder disorders and can provide an objective basis for the diagnosis, classification and identification of sleep disorders.
Flinders Fatigue Scale | baseline; 4 weeks; 12weeks
  The Flinders Fatigue Scale is a 7-item scale that measures various characteristics of fatigue. Total fatigue scores range from 0 to 31, with higher scores indicating more severe fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Healthcare Hospital, Changsha, Hunan, China